CLINICAL TRIAL: NCT02174497
Title: One-Day Bowel Preparation With Polyethylene Glycol 3350 (Miralax®) is as Effective and Safe as Three-Day Preparation for Colonoscopy in Children
Brief Title: One-Day Versus Three-Day Bowel Preparation for Colonoscopy in Children
Status: Completed | Type: Observational
Sponsor: St. John Health System, Michigan (Other)
Responsible Party: Principal Investigator, Hernando Lyons, MD, Clinical Assistant Professor of Pediatrics, St. John Health System, Michigan
Other Study IDs: OMB No 0925-0586
Record Dates: First submitted 2014-05-21; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Bowel Preparation; Pediatric Colonoscopy
Keywords: Pediatric Colonoscopy; Bowel Preparation; Safety; Tolerability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: Three day Bowel Preparation
- Study Arm: One day Bowel Preparation

SUMMARY:
This was a blinded study conducted on the efficacy and safety of a one-day versus a three-day bowel preparation in a pediatric population. Limited data is available in this regard, and this study supports the use of a one-day bowel preparation, as this is both safe and effective.

DETAILED DESCRIPTION:
Colonoscopy in children and young adults is performed by gastroenterologists for a variety of indications, including but not limited to evaluation of rectal bleeding, chronic diarrhea, family history of polyposis syndromes and surveillance for colon cancer in patients with inflammatory bowel disease. A successful bowel preparation that enables clear visualization of the intestinal mucosa is essential to diagnose and treat the underlying pathology. Currently, gastroenterologists use a variety of colon cleansing preparations, but Polyethylene Glycol (PEG) 3350 given for three to four days appears to be standard. Though it is well tolerated, safe and effective the duration of preparation may cause disruption to the routine and missed school days. To date, there is limited data that shows efficacy of a shorter duration of bowel preparation with PEG. This study aims to compare the efficacy and safety of a one-day preparation with that of a three-day preparation with PEG 3350 as preparation for colonoscopy in children and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Patients referred for an outpatient colonoscopy

Exclusion Criteria:

* None

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children between 2 and 21 years of age undergoing elective colonoscopy were enrolled into the study.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2008-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety of a one day versus a three day colonoscopy preparation in a pediatric population | 02/08-06/10 (28 months)
  The Safety of the different preparations was documented by monitoring serum electrolytes before and after the preparation.

SECONDARY OUTCOMES:
Tolerability of a one day versus a three day colonoscopy preparation in a pediatric population | 02/08-06/10 (28 months)
  The tolerability was documented by monitoring the patient's clinical ability to consume the entire colonoscopy preparation without abdominal pain, nausea or vomiting. Furthermore, this was objectively documented by monitoring and recording the following parameters: Ease of Administration, Compliance, Willingness to take again

CONTACTS AND LOCATIONS:
Locations (1):
- St. John Hospital and Medical Center, Detroit, Michigan, United States

REFERENCES:
- [Derived] Sorser SA, Konanki V, Hursh A, Hagglund K, Lyons H. 1-day bowel preparation with polyethylene glycol 3350 is as effective and safe as a 3-day preparation for colonoscopy in children. BMC Res Notes. 2014 Sep 15;7:648. doi: 10.1186/1756-0500-7-648. PMID 25223547